CLINICAL TRIAL: NCT03440034
Title: An Open-Label Pilot Study of Pioglitazone in Sporadic Inclusion Body Myositis
Brief Title: Study of Pioglitazone in Sporadic Inclusion Body Myositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00130996
Record Dates: First submitted 2017-11-14; First posted 2018-02-20 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-08

CONDITIONS: Myositis; Inclusion Body Myositis; Muscular Diseases; Musculoskeletal Disease; Neuromuscular Diseases; Nervous System Diseases
Keywords: IBM; inclusion body myositis
MeSH Terms: conditions — Myositis; Myositis, Inclusion Body; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized trial in 15 patients with sIBM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pioglitazone (Experimental): All subjects will be provided Pioglitazone 15mg tablets, total dose of 45mg (3 tablets) for oral administration once daily. 32-week treatment period.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone comes as a tablet to take by mouth and can be taken with or without food.
  Other Names: Actos

SUMMARY:
A study looking at the effect of pioglitazone in skeletal muscle of patients with sporadic inclusion body myositis (sIBM).

DETAILED DESCRIPTION:
This is a 52-week, Phase 1, open-label, single center, proof of concept study of FDA-approved pioglitazone in adult patients with sporadic inclusion body myositis (sIBM). The trial consists of a 4-week screening period;16-week "lead-in" period during which all subjects are observed off-treatment. At Week 16, all subjects will be started on pioglitazone at a dose of 30 mg daily. The dose will be uptitrated to a goal dose of 45 mg daily after 2 weeks; 32-week treatment period with all subjects on 45 mg daily dose of pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosis of sporadic inclusion body myositis (sIBM) based on the sIBM Diagnostic Criteria established by the 2010 European Neuromuscular Center.
* Must be able to ambulate at least 20 feet, with or without the use of an assistive device. Patients may not use another person, wall, or furniture for support.
* Must be able to rise from a chair without support from another person or device.
* Premenopausal women must have a negative serum pregnancy test prior to dosing with study medication.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* A history of diabetes mellitus, or prior or concurrent treatment with any diabetes therapy
* Use of chronic immunosuppressive therapy including corticosteroids or intravenous immune globulin (IVIG) within the past 6 months.
* Use of Vitamin E supplements within the past 3 months
* Creatine kinase (CK) > 15x the upper limit of normal
* Any condition other than sIBM that causes significant muscle pain, muscle weakness, muscle atrophy, or joint pain. This includes but is not limited to such neurologic and neuromuscular diseases as polymyositis or dermatomyositis, myasthenia gravis, amyotrophic lateral sclerosis, stroke, multiple sclerosis, epilepsy, muscular dystrophy, fibromyalgia, rheumatoid arthritis, spinal cord injury or degenerative disease of the spine. Osteoarthritis is not exclusionary unless it limits the patient's ability to comply with study tasks. Patients with a history of a hip or vertebral fracture within the past year or surgical hip or knee replacement within the past six months will be excluded.
* Patients receiving any medications or substances that are inhibitors or inducers of CYP2C8 are ineligible. These medications include but are not limited to Gemfibrozil, Rifampin, and warfarin.
* Pregnant women
* History of cancer less than five years prior, other than local basal or squamous cell cancer.
* Patient has any medical condition or laboratory finding during screening, which, in the investigator's opinion may interfere with participation, confound the results, or pose any additional risk to the patient.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Peroxisome proliferator-activated receptor gamma coactivator 1-alpha target gene expression | 4 weeks, 16 weeks, 32 weeks after baseline
  Effect of 45 milligram pioglitazone dose on the expression of Peroxisome proliferator-activated receptor gamma coactivator 1-alpha target genes

CONTACTS AND LOCATIONS:
Overall Officials: Jemima Albayda, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No